CLINICAL TRIAL: NCT03992404
Title: Prospective, Randomized, Double-blind, Placebo-controlled, Multicenter Study to Investigate the Efficacy and Safety of NT 201 in the Treatment of Lower Limb Spasticity Caused by Stroke or Traumatic Brain Injury in Adult Subjects, Followed by an Open Label Extension With or Without Combined Upper Limb Treatment
Brief Title: Study to Compare the Efficacy and Safety of NT 201 (Botulinum Toxin) With Placebo for the Treatment of Lower Limb Spasticity Caused by Stroke or Traumatic Brain Injury
Acronym: PATTERN
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Merz Pharmaceuticals GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M602011014; 2018-001639-35 (EudraCT Number)
Record Dates: First submitted 2019-06-18; First posted 2019-06-20 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Lower Limb or Combined Lower Limb and Upper Limb Spasticity Due to Stroke or Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — incobotulinumtoxinA; Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NT 201 (IncobotulinumtoxinA, Xeomin) (Experimental): Main Period (1 treatment cycle): subjects to receive intramuscular injection of NT 201 (400 units) into muscles of the lower limb.
  Open Label Extension Period (4-5 treatment cycles): subjects to receive intramuscular injection of NT 201 (up to 800 units) into muscles of the lower limb and upper limb, if indicated.
  Interventions: Drug: NT 201
- Placebo (Placebo Comparator): Main Period (1 treatment cycle): subjects to receive intramuscular placebo injection into muscles of the lower limb.
  Open Label Extension Period (4-5 treatment cycles): subjects to receive intramuscular injection of NT 201 (up to 800 units) into muscles of the lower limb and upper limb, if indicated.
  Interventions: Drug: NT 201; Drug: Placebo

INTERVENTIONS:
Drug: NT 201 — Active ingredient: Clostridium Botulinum neurotoxin Type A free from complexing proteins. Solution for injection prepared by reconstitution of powder with 0.9% Sodium Chloride (NaCl).
  Other Names: IncobotulinumtoxinA; Incobotulinumtoxin A; Xeomin; Botulinum toxin type A (150 kiloDalton), free from complexing proteins
Drug: Placebo — Solution for injection prepared by reconstitution of powder with 0.9% Sodium Chloride (NaCl).
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether a single treatment with administration of 400 Units NT 201 (botulinum toxin) is superior to placebo (no medicine) for the treatment of lower limb spasticity caused by stroke or traumatic brain injury (Main Period). Participants will be assigned to the treatment groups by chance and neither the participants nor the research staff who interact with them will know the allocation.

The following 4 to 5 treatment cycles will investigate the safety and tolerability of treatment with NT 201 (botulinum toxin) when administered in doses between 400 and 800 Units (Open Label Extension Period). All participants will receive the treatment and the dose will depend on whether only lower limb spasticity or combined upper and lower limb spasticity are treated.

ELIGIBILITY:
Inclusion Criteria:

* Female or male subject ≥ 18 years and ≤ 85 years at screening
* Diagnosis of lower limb spasticity with or without upper limb spasticity of the same body side caused by stroke or traumatic brain injury
* Disabling ankle flexor spasticity presenting as pes equinus or pes equinovarus
* Modified Ashworth Scale-Bohannon [MAS] score of 2 or 3 points in the ankle plantar flexor of the target lower limb (supine position, knee extended)
* Minimum passive range of motion in ankle of the target lower limb (supine position, knee extended): 10°dorsiflexion and 20°plantarflexion
* At least 4 months since last botulinum neurotoxin [BoNT] injection for treatment of spasticity or any other condition
* For subjects receiving anticoagulation therapy, the investigator confirms and documents that the subject has an:
* Activated partial thromboplastin time [aPTT] ≤ 80 seconds (subjects on dabigatran or other direct thrombin inhibitors) or
* International normalized ratio [INR] value of ≤ 2.5 (subjects on coumarins or other anticoagulants monitored by INR)

Exclusion Criteria:

* Generalized disorders of muscle activity (e.g. myasthenia gravis, Lambert Eaton syndrome, amyotrophic lateral sclerosis) or any other significant peripheral neuromuscular dysfunction which might interfere with the study
* Bilateral lower limb paresis/paralysis/spasticity or tetraparesis/paralysis/spasticity
* Body weight < 50 kg
* Severe atrophy of the target limb muscles
* Previous, ongoing or planned treatments of spasticity with intrathecal baclofen
* Previous, ongoing, or planned treatments of spasticity in the target lower limb with any of the following procedures: Surgical Intervention; Alcohol or phenol block; Muscle afferent block
* Physiotherapy or use of orthoses or splints at the target limb initiated less than 4 weeks before screening or expected to change during the double blind phase of the study
* Current or planned treatment with parenterally administered drugs that interfere with neuromuscular transmission (e.g. intrathecal baclofen, tubocurarine type muscle relaxants used in anesthesia), or local anesthetics in the treated region within 2 weeks prior to screening
* Infection or inflammation at the injection sites
* Subjects with presence or history of aspiration pneumonia, recurrent lower respiratory tract infections, or compromised respiratory function as per investigator's clinical judgment
* Pregnancy (as verified by a positive pregnancy test) or breast feeding

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 603 (Actual)
Dates: Start 2019-09-16 (Actual); Primary Completion 2025-06-19 (Actual); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in derived Modified Ashworth Scale-Bohannon (MAS) ankle score (knee extended) at weeks 4 to 6 | Baseline to week 4-6
  The MAS is a 6-grade scale
Co-Primary: Global Impression of Change Scale (GICS) assessed by physician at Week 4 to 6 | Week 4-6
  The GICS s a 9-grade scale
Occurrence of treatment emergent adverse events [TEAEs] in the Main Period | Baseline to week 12

SECONDARY OUTCOMES:
Change from Study Baseline in Goal Attainment Scale [GAS] at Week 6 | Baseline to week 6
  The GAS is a 6-grade scale
Global Impression of Change Scale (GICS) assessed by the study subject at Week 4 to 6 | Week 4-6
  The GICS s a 9-grade scale
Global Impression of Change Scale (GICS) assessed by the caregiver at Week 4 to 6 | Week 4-6
  The GICS s a 9-grade scale

CONTACTS AND LOCATIONS:
Overall Officials: Merz Medical Expert, Study Director — Merz Pharmaceuticals GmbH
Locations (71):
- United States (15):
  - Physical Medicine and Rehabilitation at University of Alabama at Birmingham; Merz investigational site #0010479, Birmingham, Alabama
  - University of Arkansas for Medical Sciences, Merz investigational site #0010481, Little Rock, Arkansas
  - Rancho Research Institute at Rancho Los Amigos National Rehabilitation Center; Merz investigational site #0010184, Downey, California
  - New England institute for clinical research; Merz Investigational Site #0010441, Stamford, Connecticut
  - Nova Clinical Research, Merz investigational site #0010474, Brandenton, Florida
  - Brooks Rehabilitation Clinical Integration and Research, Merz investigational site #0010483, Jacksonville, Florida
  - Sarasota Memorial Health Care System, Rehabilitation Medicine, Merz investigational site #0010478, Sarasota, Florida
  - Neurology Center of New England P.C., Merz investigative site #0010476, Foxborough, Massachusetts
  - Howard A. Rusk Rehabilitation Center; Merz investigational site #0010283, Columbia, Missouri
  - Icahn School of Medicine at Mount Sinai, Neurology Department, Merz Investigational Site #0010191, New York, New York
  - Weill Cornell Medical Center, Department of Rehabilitation Medicine; Merz Investigational Site #0010440, New York, New York
  - University of Pittsburgh Medical Center, Physical Medicine & Rehabiliation, Merz Investigational Site #0010211, Pittsburgh, Pennsylvania
  - UT Southwestern Medical Center, Department of Physical Medicine & Rehabilitation, Merz investigational site #0010082, Dallas, Texas
  - University of Texas Health Science Center McGovern, Medical School Department of PM&R; merz investigational site #0010183, Houston, Texas
  - Medical College of Wisconsin,Department of PM&R, Merz Investigational Site #0010237, Milwaukee, Wisconsin
- Belgium (4):
  - CHU Brugmann Neurology; Merz investigational site #0320015, Brussels
  - UCL Bruxelles, Physical Medicine & Rehabilitation Department, Merz Investigational Site #0320013, Brussels
  - UZ Leuven Pellenberg campus; Merz investigational site #0320014, Pellenberg
  - UCL Mont Godinne, Physical Medicine & Rehabilitation Department; Merz Investigational Site #0320008, Yvoir
- Glenrose Rehabilitation Hospital, Merz investigational site #0010195, Edmonton, Canada
- Czechia (3):
  - Neurology and Physiotherapy Skopalikova, Merz Investigational Site #4200049, Brno
  - University Hospital Ostrava; Neurology Departement, Merz investigational site #4200024, Ostrava
  - Pardubice Regional Hospital; Merz investigational site #4200025, Pardubice
- France (5):
  - Raymond Poincaré University Hospital, Service de MPR Pôle Handicap-Rééducation, Merz Investigational site #00330018, Garches
  - CHU Lille/Hôpital Swynghedauw; investigational site # 0330045, Lille
  - Pôle Saint-Hélier; Merz investigational site #0330024, Rennes
  - Institut Universitaire de Readaptation Clemenceau, Physical Medicine / Rehabilitation Medecine, Merz Investigational site # 0330063, Strasbourg
  - Rangueil Hospital-University Hospital Center (CHU) of Toulouse, Médecine physique et de réadaptation, Merz investigational site #0330025, Toulouse
- Germany (7):
  - Uniklinik RWTH Aachen, Neurologie, Merz Investigational Site #0490191, Aachen
  - Neurologie Bewegt; Merz Investigational site #0490378, Berlin
  - University of Bonn Medical Center, Department of Neurodegenerative disease, Merz investigational site #0490390, Bonn
  - Heinrich Heine University Duesseldorf, Department of Neurology; Merz Investigational Site #0490071, Düsseldorf
  - Universitätsklinikum Hamburg-Eppendorf, Merz Investigational site #0490079, Hamburg
  - DKD HELIOS Medical Center, Fachbereich Neurologie, Merz Investigational Site #0490081, Wiesbaden
  - Neurologische Klinik und Poliklinik des Universitätsklinikums Würzburg, Merz Investigational Site #0490302, Würzburg
- Hungary (3):
  - Petz Hospital, Neurology, Merz Investigational Site #0360010, Győr
  - St.Damjan Hospital, Kisvarda; Merz investigational site #0360019, Kisvárda
  - University of Szeged, Department of Neurology, Merz investigational site #0360008, Szeged
- Italy (4):
  - Azienda Ospedaliera Universitaria Ospedali Riuniti Di Foggia; Merz Investigational Site #0390018, Foggia
  - IRCCS Ospedale Policlinico S. Martino, U.O.Complessa Riabilitazione e Rieducazione Funzionale; Merz investigational site #0390020, Genova
  - Ospedale Maggiore della Carita, Dipartimento di Medicina fisica e Riabilitativa, Merz Investigational Site #0390017, Novara
  - Ospedale Alfredo Fiorini, UOSD Neurologia Universitaria; Merz Investigational site #0390022, Terracina
- Poland (9):
  - Specjalistyczna Praktyka Lekarska Dr. n. med Stanisław Ochudło, Merz Investigational Site #0480077, Katowice
  - Specjalistyczne Gabinety Sp z o.o., Merz Investigational Site #0480059, Krakow
  - NeuroKlinika Gabinet Lekarski Prof Andrzej Bogucki, Merz Investigational Site #0480101, Lodz
  - Indywidualna Praktyka Lekarska dr. hab. Med. Anna Szczepanska-Szerej, Merz Investigational Site #0480096, Lublin
  - Filia 7 Centrum Kompleksowej Rehabilitacji Sp. z o.o., Merz Investigational Site #0480100, Warsaw
  - Projekt Samodzielni Sp z o.o., Merz Investigational Site #0480099, Warsaw
  - Instytut Psychiatrii i Neurologii, II Klinika Neurologiczna, Merz Investigational Site #0480023, Warsaw
  - Mazowiecki Szpital Brodnowski, Merz investigational site #0480064, Warsaw
  - Neuryt Diagnostyka I Terapia Neurologiczna, Merz investigational site #0480106, Wroclaw
- Russia (4):
  - Federal State Budgetary Educational Institution of Higher Education "Krasnoyarsk State Medical University n.a. Professor V.F. Voino-Yasenetskiy of Ministry Healthcare of Russian Federation", Merz Investigational Site #0070306, Krasnoyarsk
  - State Autonomous Institution of Healthcare of Moscow City "Moscow Scientific and Practical Centre of Medical Rehabilitation, Regenerative and Sports Medicine of Moscow City Healthcare Department", Merz Investigational Site #0070011, Moscow
  - Federal State Autonomous Institution "National Medical Research Centre "Treatment and Rehabilitation" of the Ministry of Health of the Russian Federation, Neurology department, Merz Investigational Site # 0070305, Moscow
  - Federal State Budgetary Institution "National Medical Research Centre of Psychiatry and Neurology n.a. V.M. Bekhterev" of the Ministry of Healthcare of the Russian Federation, Merz Investigational Site #0070009, Saint Petersburg
- Slovakia (2):
  - University Hospital Bratislav, 2nd Dept. of Neurology, Merz Investigational Site # 4210005, Bratislava
  - Neurologicka klinika, Fakultna nemocnica Trnava; Merz investigational site #4210009, Trnava
- Spain (3):
  - Hospital Universitario Juan Ramón Jiménez, Merz Investigational Site #0340037, Huelva
  - Hospital Universitario La Paz, Merz Investigational Site #0340007, Madrid
  - Hospital Universitari Mútua de Terrassa, Merz Investigational Site #0340003, Terrassa
- Switzerland (3):
  - University Hospital of Bern, Center of Parkinson's diseases and Movement disorders (ZfPB), Merz investigational site #0410015, Bern
  - HFR Fribourg - Hôpital Cantonal, Department of Rehabilitation, Merz Investigational site #0410014, Meyriez
  - CRR, Mee Suva (Clinique romande de réadaptation), Merz investigational site #0410016, Sion
- Ukraine (5):
  - Institute of Neurology, Psychiatry and Narcology of NAMS of Ukraine, MC "Neuron", Merz Investigational Site #3800018, Kharkiv
  - Institute of Neurology, Psychiatry and Narcology of NAMS of Ukraine; Merz Investigational Site #3800019, Kharkiv
  - Lviv regional clinical hospital; Merz investigational site # 3800020, Lviv
  - Rivne City Hospital 2, Department of Clinical Neurology and Neurorehabilitation; Merz investigational site #3800016, Rivne
  - NPE "Regional Clinical Centre of Neurosurgery and Neurology" Transcarpathian Regional Council; Merz investigational site #3800014, Uzhhorod
- United Kingdom (3):
  - Cambridge University Hospitals NHS Foundation Trust; Merz Investigational Site 0440023, Cambridge
  - Royal Devon and Exeter Foundation Trust Hospital, Department of Neurology, Merz Investigational Site #0440047, Exeter
  - The Walton Centre NHS Foundation Trust; Neuroscience Research Centre; Merz Investigational site #0440004, Liverpool

IPD SHARING:
Plan to Share IPD: No